CLINICAL TRIAL: NCT00297258
Title: Phase II Study of GW786034 in Patients With Relapsed or Refractory Soft Tissue Sarcoma
Brief Title: Pazopanib In Patients With Relapsed Or Refractory Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG20002; NCT00293449 (obsolete NCT alias)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma; Synovial sarcoma; Pazopanib(GW786034); Adipocytic tumors; Leiomyosarcoma; Phase II
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial; Leiomyosarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pazopanib — oral tablet
  Other Names: GW786034

SUMMARY:
The purpose of this study is to evaluate the activity and tolerability of pazopanib in subjects with advanced and/or metastatic soft tissue sarcoma who have relapsed following standard therapies or for whom no standard therapy exists and to characterize the pharmacokinetics of pazopanib in this subject population.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of high or intermediate grade malignant soft tissue sarcoma, or cytological evidence in case of presence of multiple metastases. List of eligible and ineligible tumours are included in the protocol.
* Formalin fixed paraffin embedded tumour blocks and representative H/E (haematoxylin/eosin) slides must be available for histological central review. Histological central review is not required before treatment start but is mandatory within 3 months of registration. Local histopathological diagnosis will be accepted for entry into the study.
* Presence of measurable disease (according to RECIST criteria).
* Relapsed or refractory disease incurable by surgery or radiotherapy.
* Evidence of objective progression within the last 6 months (RECIST) documented by measurements of disease,
* Patients must either not be eligible for chemotherapy (for instance because of age, or because of a biological condition, or because of patient-refusal) or must have received no more than one combination or two single agents chemotherapy regimen for advanced disease; (neo) adjuvant therapy is not counted towards this requirement.
* At least 18 years of age
* WHO performance status 0 or 1
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function
* PT / PTT less than 1.2 x UNL.
* LVEF above the lower limit of normal for the institution, based on ECHO or MUGA
* Able to swallow and retain oral medication
* Women should not be of childbearing potential and agree to use contraceptive methods (Oral contraceptives are not allowed).
* Absence of any serious and/or unstable pre-existing medical, psychiatric or other condition (including lab abnormality) that could interfere with patient safety or obtaining informed consent.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed with the patient before registration in the trial.
* Written informed consent is given according to ICH/GCP, and national/local regulations before patient registration/randomization.

Exclusion Criteria:

* history of leptomeningeal or brain metastases
* history of malignancies other than sarcoma (except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or the patient has been free of any other malignancies for greater than 3 years).
* Class II, III or IV heart failure (NYHA classification). A patient who has a history of class II heart failure and is asymptomatic on treatment may be considered eligible.
* Arterial or venous thrombosis, myocardial infarction, unstable angina, cardiac angioplasty or stenting within the last 3 months
* Uncontrolled or poorly controlled hypertension. Initiation or adjustment of BP medications is permitted prior to study entry, provided that patient has 3 consecutive BP readings less than 150 / 90 mm Hg each separated by a minimum of 24 hrs. These readings need to be collected prior to registration in the study.
* Women of childbearing potential, who are pregnant (negative serum pregnancy test at entry) or lactating.
* Therapeutic dose warfarin. Low molecular weight heparin and prophylactic low dose warfarin are permitted. PT/INR and PPT must meet the above inclusion criteria.
* Concurrent therapy with any specifically prohibited medication or requirement for using any of these medications during treatment with pazopanib
* Major surgery, hormonal therapy (other than replacement), chemotherapy or radiotherapy, immunotherapy or other investigational agent within the last 28 days and/or not recovered from prior therapy within the last 28 days. Use of erythropoietin is considered supportive care and is permitted. The patient should have recovered from prior surgery and have no open wounds.
* History of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption, distribution, metabolism or excretion of study drugs. No unresolved bowel obstruction or diarrhea.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- France (4):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Budapest, Hungary
- Netherlands (3):
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Rotterdam
- United Kingdom (6):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Background] Sleijfer S, Ray-Coquard I, Papai Z, Le Cesne A, Scurr M, Schoffski P, Collin F, Pandite L, Marreaud S, De Brauwer A, van Glabbeke M, Verweij J, Blay JY. Pazopanib, a multikinase angiogenesis inhibitor, in patients with relapsed or refractory advanced soft tissue sarcoma: a phase II study from the European organisation for research and treatment of cancer-soft tissue and bone sarcoma group (EORTC study 62043). J Clin Oncol. 2009 Jul 1;27(19):3126-32. doi: 10.1200/JCO.2008.21.3223. Epub 2009 May 18. PMID 19451427
- [Background] Sleijfer S, Gorlia T, Lamers C, Burger H, Blay JY, Le Cesne A, Scurr M, Collin F, Pandite L, Marreaud S, Hohenberger P. Cytokine and angiogenic factors associated with efficacy and toxicity of pazopanib in advanced soft-tissue sarcoma: an EORTC-STBSG study. Br J Cancer. 2012 Aug 7;107(4):639-45. doi: 10.1038/bjc.2012.328. Epub 2012 Jul 17. PMID 22805326
- [Derived] Kasper B, Sleijfer S, Litiere S, Marreaud S, Verweij J, Hodge RA, Bauer S, Kerst JM, van der Graaf WTA. Long-term responders and survivors on pazopanib for advanced soft tissue sarcomas: subanalysis of two European Organisation for Research and Treatment of Cancer (EORTC) clinical trials 62043 and 62072. Ann Oncol. 2014 Mar;25(3):719-724. doi: 10.1093/annonc/mdt586. Epub 2014 Feb 6. PMID 24504442

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib 800 mg: Pazopanib 800 milligram (mg) (tablets) administered orally once a day
Period: Overall Study
Arm/Group | Pazopanib 800 mg
Started | 142
Completed | 0
Not Completed | 142
Not completed — Disease Progression, Relapse, Death | 120
Not completed — Toxicity (or Toxic Death) | 10
Not completed — Patient Refusal: Not Related to Toxicity | 2
Not completed — Intercurrent Illness | 3
Not completed — Intercurrent Death | 2
Not completed — Deteriorization of General Condition | 1
Not completed — Radiotherapy to Destroy Last Lesion | 1
Not completed — Surgery Performed on Target Lesion | 1
Not completed — Switch to Commercial Treatment | 1
Not completed — Interruption: Cold/Flu-like Symptoms | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 142
Age, Continuous [Median (Full Range); unit: years] — Includes all participants enrolled in the study
  years | 51.0 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 71

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at Week 12
Description: Progression free survival at week 12 is the number of participants who had a complete response (CR, all detectable tumor had disappeared) or a partial response (PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum) or stable disease (SD, no change) 12 weeks from start of therapy, per response evaluation criteria in solid tumors (RECIST v1.0). Clinical progression is progression of disease without documented radiological evidence. Progressive disease (PD), a >=20% increase in target lesions.
Time Frame: Week 12
Population: Intent-to-Treat (ITT) Population: All eligible participants entered into the study and who had taken >=1 dose of investigational product. Four participants were considered not evaluable for efficacy by the study coordinator for one of the following reasons: absence of target lesions, documented progression at trial entry, or ineligible histology.
Measure: Number; unit: participants
Groups:
- Pazopanib 800 mg - Adipocytic Tumors; Pazopanib 800 mg - Leiomyosarcoma; Pazopanib 800 mg - Synovial Sarcoma; Pazopanib 800mg - Other Soft Tissue Sarcoma (STS): Pazopanib 800 mg (tablets) administered orally once a day
Arm/Group | Pazopanib 800 mg - Adipocytic Tumors | Pazopanib 800 mg - Leiomyosarcoma | Pazopanib 800 mg - Synovial Sarcoma | Pazopanib 800mg - Other Soft Tissue Sarcoma (STS)
Number analyzed (Participants) | 19 | 41 | 37 | 41
participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 4 | 1
  Stable Disease | 5 | 16 | 14 | 16
  Progressive Disease | 13 | 19 | 15 | 21
  Unknown | 0 | 2 | 0 | 1
  Missing | 1 | 3 | 4 | 2
  CR+PR+SD | 5 | 17 | 18 | 17
Statistical Analysis 1: Comparison: Pazopanib 800 mg - Adipocytic Tumors; Test type: Superiority or Other; p = 0.653, binomial exact method; percentage of participants = 46, 90% CI [11.0 to 47.6] — The estimated value represents the percentage of participants with a CR, a PR, or SD
Statistical Analysis 2: Comparison: Pazopanib 800 mg - Leiomyosarcoma; Test type: Superiority or Other; p = 0.003, binomial exact method; percentage of participants = 41, 90% CI [28.4 to 55.5] — The estimated value represents the percentage of participants with a CR, a PR, or SD
Statistical Analysis 3: Comparison: Pazopanib 800 mg - Synovial Sarcoma; Test type: Superiority or Other; p < 0.001, binomial exact method; percentage of participants = 49, 90% CI [34.3 to 63.2] — The estimated value represents the percentage of participants with a CR, a PR, or SD
Statistical Analysis 4: Comparison: Pazopanib 800mg - Other Soft Tissue Sarcoma (STS); Test type: Superiority or Other; p = 0.003, binomial exact method; percentage of participants = 41, 90% CI [28.4 to 55.5] — The estimated value represents the percentage of participants with a CR, a PR, or SD

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from start of therapy until death. Participants who were still alive at the time of analysis were censored.
Time Frame: Start of therapy until death (up to approximately 5 years)
Population: ITT Population. Four participants were considered not evaluable for efficacy by the study coordinator for one of the following reasons: absence of target lesions, documented progression at trial entry, or ineligible histology.
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Pazopanib 800 mg - Adipocytic Tumors | Pazopanib 800 mg - Leiomyosarcoma | Pazopanib 800 mg - Synovial Sarcoma | Pazopanib 800mg - Other Soft Tissue Sarcoma (STS)
Number analyzed (Participants) | 19 | 41 | 37 | 41
years | 28.1 [18.3 to 84.0] | 50.9 [46.1 to 76.4] | 44.6 [33.0 to 57.6] | 42.6 [33.1 to 49.3]

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the interval between the start of treatment and the earliest date of disease progression or death due to any cause. Assessments of progression were made by the investigator.
Time Frame: Start of therapy until progression (up to approximately 5 years)
Population: Intent-to-Treat (ITT) Population: all eligible participants who had started therapy. Four participants were considered not evaluable for efficacy by the study coordinator for one of the following reasons: absence of target lesions, documented progression at trial entry, or ineligible histology.
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Pazopanib 800 mg - Adipocytic Tumors | Pazopanib 800 mg - Leiomyosarcoma | Pazopanib 800 mg - Synovial Sarcoma | Pazopanib 800mg - Other Soft Tissue Sarcoma (STS)
Number analyzed (Participants) | 19 | 41 | 37 | 41
years | 11.1 [7.1 to 11.9] | 17.2 [12.0 to 24.1] | 23.4 [11.7 to 29.3] | 14.0 [12.0 to 36.3]

4. Secondary Outcome: Overall Response
Description: Overall response is the number of participants who had a best outcome of a complete response (CR, all detectable tumor had disappeared) or a partial response (PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum) per response evaluation criteria in solid tumors (RECIST v1.0) at some point during the study. Progressive disease (PD), a >=20% increase in target lesions. Clinical progression is progression of disease without documented radiological evidence.
Time Frame: Baseline until either response or progression (up to approximately 5 years)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg - Adipocytic Tumors | Pazopanib 800 mg - Leiomyosarcoma | Pazopanib 800 mg - Synovial Sarcoma | Pazopanib 800mg - Other Soft Tissue Sarcoma (STS)
Number analyzed (Participants) | 19 | 41 | 37 | 41
participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 4 | 3
  Stable Disease | 5 | 17 | 14 | 14
  Progressive Disease | 13 | 19 | 13 | 21
  Unknown | 1 | 4 | 6 | 3
  Missing | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Entire Study (average of 8.24 years).
Arm/Group | Pazopanib 800 mg
Serious Adverse Events (participants affected / at risk) | 39/142
Other Adverse Events (participants affected / at risk) | 137/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=142)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Ileal perforation (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 2
Chest pain (General disorders) | 2
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Oedema (General disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 5
Hypertension (Vascular disorders) | 3
Pnuemonia (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Vision blurred (Eye disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=142)
Fatigue (General disorders) | 84
Diarrhoea (Gastrointestinal disorders) | 62
Nausea (Gastrointestinal disorders) | 60
Hypertension (Vascular disorders) | 57
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 53
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 51
Vomiting (Gastrointestinal disorders) | 48
Decreased appetite (Metabolism and nutrition disorders) | 45
Weight decreased (Metabolism and nutrition disorders) | 45
Constipation (Gastrointestinal disorders) | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 33
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31
Headache (Nervous system disorders) | 30
Abdominal pain (Gastrointestinal disorders) | 27
Exfoliative rash (Skin and subcutaneous tissue disorders) | 23
Oedema (General disorders) | 21
Stomatitis (Gastrointestinal disorders) | 18
Chest pain (General disorders) | 17
Abdominal pain upper (Gastrointestinal disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 15
Pyrexia (General disorders) | 17
Dysgeusia (Nervous system disorders) | 13
Abdominal distension (Gastrointestinal disorders) | 12
Anxiety (Psychiatric disorders) | 13
Dizziness (Nervous system disorders) | 12
Insomnia (Psychiatric disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.